CLINICAL TRIAL: NCT01946217
Title: Improving Participation in AMC Clinical Trials (IMPACTS)
Brief Title: Factors Affecting Patient Participation in AIDS Malignancy Clinical Trials Consortium Clinical Trials
Status: Completed | Type: Observational
Sponsor: AIDS Malignancy Consortium (Network)
Collaborators: National Cancer Institute (NCI) (NIH); The Emmes Company, LLC (Industry); University of Arkansas (Other)
Responsible Party: Sponsor
Other Study IDs: AMC-S006; NCI-2013-01152 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); AMC-S006 (Other: AIDS - Associated Malignancies Clinical Trials Consortium); AMC-S006 (Other: CTEP); U01CA121947 (NIH)
Record Dates: First submitted 2013-09-17; First posted 2013-09-19 (Estimated); Last update posted 2016-08-18 (Estimated); Status verified 2016-08

CONDITIONS: HIV Infection; Malignant Neoplasm; Precancerous Condition
MeSH Terms: conditions — HIV Infections; Neoplasms; Precancerous Conditions

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Observational (questionnaire administration): Participants complete the IMPACTS survey comprising questions about socio-demographic information and clinical trial participation.
  Interventions: Other: questionnaire administration

INTERVENTIONS:
Other: questionnaire administration — Ancillary studies

SUMMARY:
This pilot research trial studies factors affecting patient participation in Acquired Immune Deficiency Syndrome (AIDS) Malignancy Clinical Trials Consortium clinical trials. Determining how patients makes decisions about participating in a clinical trial may help doctors plan clinical trials in which more patients are willing to participate and are satisfied with their decision to participate.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To identify participant-level factors affecting recruitment of potentially eligible participants in AIDS Malignancy Clinical Trials Consortium (AMC) studies at core and affiliated sites.

SECONDARY OBJECTIVES:

I. To describe the socio-demographic characteristics for participation and non-participation in AMC clinical trials among all approached volunteers across AMC sites.

II. To characterize socio-demographic characteristics with motivation and decision making among those who consented to participate in an AMC trial.

III. To identify the perceived barriers associated with clinical trial participation among those who did not consent to participate in an AMC clinical trial.

IV. To better understand how potential study volunteers learn about AMC clinical trials and by what means are they referred to a particular study.

OUTLINE:

Participants complete the Improving Participation in AMC Clinical Trials (IMPACTS) survey comprising questions about socio-demographic information and clinical trial participation.

ELIGIBILITY:
Inclusion Criteria:

* HIV-infected participants
* Cancer or anal dysplasia diagnosis
* Offered informed consent on an AMC interventional clinical trial
* Ability to understand and the willingness to sign a written informed consent document

Exclusion Criteria:

* Inability to provide informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: HIV-infected persons with a diagnosis of anal dysplasia or cancer who are offered informed consent on an AMC interventional clinical trial.
Sampling Method: Non-Probability Sample
Enrollment: 82 (Actual)
Dates: Start 2013-09; Primary Completion 2015-09 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
Participant level factors affecting recruitment of potentially eligible participants in AMC intervention studies | Up to 2 weeks
  The proportion of individuals who are screened and agree to enroll in a clinical trial will be estimated with the binomial proportion and its 95% confidence interval.

SECONDARY OUTCOMES:
Socio-demographic characteristics for participation and non-participation in AMC clinical trials among all approached volunteers across AMC sites | Up to 2 weeks
  Chi-square tests will be used to compare the characteristics of those who enrolled in a clinical trial with those who did not with respect to sociodemographic characteristics, sexual orientation, and disease-type and design type.
Socio-demographic characteristics with motivation and decision making among those who consented to participate in an AMC trial | Up to 2 weeks
  Chi-square tests will be used to compare the characteristics of those who enrolled in a clinical trial with those who did not with respect to sociodemographic characteristics, sexual orientation, and disease-type and design type.
Perceived barriers associated with clinical trial participation among those who did not consent to participate in an AMC clinical trial | Up to 2 weeks
  For each study participant who did not enroll in a trial, the number of barriers in each category (views and attitudes, views of other people around them, financial burden and travel) will be computed. Summary statistics (mean, standard deviation [SD], median and interquartile range) will be used to estimate number of barriers in each category. Analyses of variance will be used to assess the associations of sociodemographic characteristics, sexual orientation, disease-type and design-type with the number of barriers in each category.
Means by which volunteers are referred to a particular study | Up to 2 weeks
  For study participants who enrolled in a clinical trial, the binomial proportion will be used to estimate the proportion who answered affirmatively to each of the six statements related to decision-making about clinical trials, and the individual reasons for participating in clinical trials. For each study participant who enrolled in a trial, the number of reasons cited for participation will be computed. Summary statistics mean, SD, median and interquartile range) will be used to estimate number of reasons cited for enrollment.

CONTACTS AND LOCATIONS:
Overall Officials: Jack Burkhalter, Principal Investigator — AIDS Associated Malignancies Clinical Trials Consortium
Locations (14):
- United States (14):
  - UCLA Clinical AIDS Research and Education (CARE) Center, Los Angeles, California
  - Stroger Hospital of Cook County, Chicago, Illinois
  - Interim LSU Public Hospital, New Orleans, Louisiana
  - HIV Out-patient Clinic, New Orleans, Louisiana
  - NO AIDS Clinic, New Orleans, Louisiana
  - Laser Surgery Care, New York, New York
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - Albert Einstein Cancer Center at Albert Einstein College of Medicine, The Bronx, New York
  - Montefiore-Einstein Cancer Center, The Bronx, New York
  - Montefiore Medical Center, The Bronx, New York
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - Virginia Mason Medical Center, Seattle, Washington
  - Harborview Madison Clinic, Seattle, Washington
  - Seattle Cancer Care Alliance, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No